CLINICAL TRIAL: NCT06554886
Title: An Open Label Pilot Study Investigating the Safety and Efficacy of a Percutaneous Peripheral Cryoneurolysis Therapy in Medically Resistant Chronic Migraine
Brief Title: A Study Investigating Peripheral Cryoneurolysis in Adults With Chronic Migraine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 727678
Record Dates: First submitted 2024-06-24; First posted 2024-08-15 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Chronic Migraine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active treatment (Experimental): Cryoneurolysis
  Interventions: Device: Cryoneurolysis

INTERVENTIONS:
Device: Cryoneurolysis — Cryoneurolysis

SUMMARY:
The trial is a research study that tests a freezing technique called cryoneurolysis to see if it helps relieve pain in adults with chronic migraine. Chronic migraine is a condition that causes moderate to severe headache.

In this study, the investigators want to evaluate the freezing technique in chronic migraine. The main goal is to see how much headache relief is experienced after receiving the treatment. The investigators will also record other important information about the participants.

The study is looking to recruit 12 adults with chronic migraine to take part in the study. Participants will register their headache burden in a headache diary for at least 4 weeks before receiving treatment with the freezing technique. They will continue to register headache in the headache diary during the follow-up. After this initial treatment, participants with recurring headache can receive treatment as needed for up to two years.

The results of this study will help us decide if the freezing technique may be viable treatment option for chronic migraine and enable us plan for further studies on this treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 years at the time of signing the informed consent
2. Migraine, with or without aura, fulfilling the International Classification of Headache Disorders (ICHD) III criteria 1.3. for chronic migraine at time of inclusion, verified by a neurologist
3. History of 8 debilitating headache days per month for at least 3 consecutive months. Debilitating headache is defined as headache causing serious impairment to conduct activities of daily living despite the use of pain-relief drugs with established efficacy at the recommended dose and taken early during the attack; failure of at least two different triptans is required.
4. Chronic migraine at least for a period of 1 year prior to inclusion
5. Debut of episodic migraine before the age of 50, and chronic migraine before the age of 65.
6. The condition is pharmacologically resistant as defined in EHF guidelines as lack of efficacy, lack of tolerability and/or contraindications to at least 3 of the following drug classes

   1. Antidepressant (Amitryptyline, Venlafaxine)
   2. Antiepileptic (Topiramate or Valproate)
   3. Beta-blocker (Atenol, Metropolol, Propanolol, Timolol)
   4. Calcium channel blockers (Flunarizine or Cinnarizine)
   5. Drugs acting on the CGRP pathway (Monoclonal antibodies and gepants)
   6. Angiotensin-converting enzyme inhibitors (Lisinopril) or angiotensin II receptor blocker (Candesartan)
   7. OnabotulinumtoxinA
7. Subject has had no change in type, dosage or dose frequency of preventive headache medications < 3 months prior to baseline/screening, or a minimum of 5 half-lives, whichever is longer.
8. Subjects has not been treated with steroids orally or injections >8 weeks (excluding steroid inhalations or topical treatments) prior to baseline and agrees to refrain from steroids orally or injections during baseline and 8 weeks post-intervention.
9. Subject agrees to maintain current preventive headache medication regimens (no change in type, frequency, or dose) during baseline and 8 weeks after the intervention.
10. Be an appropriate candidate for the study intervention required in this study on the basis of the clinical judgment of the investigator
11. Capable of giving signed informed consent as which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Subject is unable to differentiate migraine from other concomitant headaches.
2. Subject with secondary headache conditions, with the exception of medication overuse headache.
3. Subject that, in the opinion of the investigator, has had no or minimal response to more than 6 adequate trials of prophylactic migraine treatment of the following drug classes:

   1. Antidepressant (Amitryptyline, Venlafaxine)
   2. Antiepileptic (Topiramate or Valproate)
   3. Beta-blocker (Atenol, Metropolol, Propanolol, Timolol)
   4. Calcium channel blockers (Flunarizine or Cinnarizine)
   5. Drugs acting on the CGRP pathway (Monoclonal antibodies and gepants)
   6. Angiotensin-converting enzyme inhibitors (Lisinopril) or angiotensin II receptor blocker (Candesartan)
   7. OnabotulinumtoxinA
4. Subject has had a change in type, dosage or dose frequency of preventive headache medications during the baseline period.
5. Ongoing abuse of drugs (including narcotics) or alcohol.
6. More than 4 days of opioid use per month (including codeine and tramadol), and any use of barbiturates
7. Other pain conditions, not intended to be treated in this study, that in the opinion of the investigator could interfere with study procedures, accurate pain reporting, and/or confound evaluation of study endpoints.
8. High probability of deterioration due to other medical conditions, that in the opinion of the investigator may confound outcome assessment.
9. Other coexisting current medical conditions, including, but not limited to, bleeding diathesis and thrombophilia, that presents excess procedural risk, in the opinion of the investigator.
10. Abnormal pain behavior, inappropriate medication use and/or unresolved psychiatric illness, that in the opinion of the investigator are significant enough to impact perception of pain, compliance with intervention and/or ability to evaluate treatment outcome.
11. Anomaly or trauma which renders the planned procedure difficult.
12. Subject currently has an active abscess or a local infection at the site of intervention based on present symptoms.
13. Subject has been diagnosed with any major infectious processes such as osteomyelitis, or primary or secondary malignancies involving skull or site of intervention that have been active or required treatment in the past 6 months.
14. Patients with any kind of conductive implant with contraindication for nerve stimulation.
15. The subject is not competent to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Headache days - severe and moderate | Weeks 5 - 8 post intervention versus baseline
  Difference in change in mean monthly headache days with moderate or severe intensity
Safety - AE and SAE | 8 weeks post-intervention
  Occurrence of treatment-emergent AE and SAE

SECONDARY OUTCOMES:
Headache days - any intensity | Weeks 5 - 8 post intervention versus baseline
  Difference in change in mean monthly headache days with any intensity
Migraine days | Weeks 5 - 8 post intervention versus baseline
  Difference in change in mean monthly migraine days
Responders 30% | Weeks 5 - 8 post-intervention
  Number of 30% responders
Responders 50% | Weeks 5 - 8 post-intervention
  Number of 50% responders
Headache Intensity | Weeks 5 - 8 post intervention versus baseline
  Difference in the mean monthly headache intensity with a 11 point VAS scale as registered in headache diary
Medication consumption | Weeks 5 - 8 post intervention versus baseline
  Difference in mean monthly days with acute medication consumption as registered in headache diary

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F Bratbak, PhD, Principal Investigator — St. Olavs Hospital
Locations (1):
- St. Olavs hospital, Trondheim, Norway